CLINICAL TRIAL: NCT04354025
Title: A Phase 2 Study of Cytokine-induced Memory-like NK Cells in Combination With Chemotherapy in Pediatric Patients With Refractory or Relapsed AML
Brief Title: Cytokine-induced Memory-like NK Cells in Combination With Chemotherapy in Pediatric Patents With Refractory or Relapsed AML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator decided not to move forward with the study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-x130
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim; Interleukin-2; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recipient: FLAG + CIML NK Cells + IL-2 (Experimental): -The recipient will begin a chemotherapy regimen of fludarabine, cytarabine and GCSF starting on Day -7. The haploidentical donor identified by HLA matching of the immediate family members will undergo non-mobilized large volume (20 L) leukapheresis on Day -1, and the NK cell product will be infused into the recipient on Day 0. CIML NK cells will be infused at maximum cell dose of 10 x 106/kg. Subcutaneous IL-2 will begin approximately 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses.
  Interventions: Biological: Cytokine induced memory-like NK cells; Drug: Fludarabine; Drug: Ara-C; Drug: G-CSF; Drug: Interleukin-2
- Donor: (Other): -On Day -1 (one day before the planned NK cell infusion), peripheral blood mononuclear cells will be collected by a single standard apheresis over 4-5 hours (with a target volume of at least 20 L) from the identified haploidentical donor. The apheresis procedure will be done as per standard institutional procedures (which may include placement of a central line if necessary). If the goal minimum NK cell dose will not be met based on the initial assessment of the leukapheresis product, a second collection/procedure may be performed.
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Biological: Cytokine induced memory-like NK cells — -The CIML NK cells (maximum dose capped at 10 x 106/kg, minimum dose allowed is 0.5 x 106/kg) will be infused on Day 0 without a filter or pump.
  Other Names: CIML NK cells
  Arms: Recipient: FLAG + CIML NK Cells + IL-2
Drug: Fludarabine — -Fludarabine (dose: 30 mg/m^2 per dose) will be given daily beginning on Day -7 for a total of 5 doses administered as an IV infusion over 30 minutes.
  Arms: Recipient: FLAG + CIML NK Cells + IL-2
Drug: Ara-C — -Ara-C (dose: 2000mg/m^2 per dose) will be given daily for a total of 5 doses administered as IV infusion over 3 hours, starting the same day as fludarabine.
  Other Names: Cytarabine
  Arms: Recipient: FLAG + CIML NK Cells + IL-2
Drug: G-CSF — -Filgrastim (dose: 5 mcg/kg per dose to a maximum of 300 mcg) will be given subcutaneously daily for a total of 5 doses starting the same day as fludarabine and ara-C.
  Other Names: Filgrastim
  Arms: Recipient: FLAG + CIML NK Cells + IL-2
Drug: Interleukin-2 — -IL-2 will be administered subcutaneously at a dose of 1 million units/m2 every other day from Day 0 to Day +12 (7 doses total).
  Other Names: IL-2
  Arms: Recipient: FLAG + CIML NK Cells + IL-2
Procedure: Leukapheresis — -Donor only
  Arms: Donor:

SUMMARY:
This phase 2 clinical trial investigates the effectiveness of cytokine-induced memory-like natural killer (CIML NK) cells in combination with FLAG chemotherapy as a treatment for refractory or relapsed AML. Previous studies in adults with AML sowed successful induction of remission and a previous phase 1 study demonstrated that CIML NK cells can be used safely in pediatric patients. This phase 2 study uses FLAG chemotherapy to lower leukemic burden and suppress the recipient's immune system to provide an optimal environment for CIML NK cell expansion and anti-leukemic activity.

ELIGIBILITY:
Inclusion Criteria:

* Refractory AML without complete remission (CR) after induction therapy (primary induction failure) or relapsed AML after obtaining a CR. Disease defined by one of the following:

  *≥ 5% blasts in the bone marrow (M2/M3 bone marrow), with or without extramedullary disease

  *absolute blast count greater than 1,000 per microliter in the peripheral blood with or without extramedullary disease.
* Age requirement for pediatric cohort: 1-21 years of age.
* Available HLA-haploidentical donor that meets the following criteria:

  * Related donor (parent, sibling, offspring, or offspring of sibling)
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus.
  * In general, good health and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
  * Negative for hepatitis, HTLV, and HIV on donor viral screen
  * Not pregnant
  * Voluntary written consent to participate in this study
* Patients with known CNS involvement with AML are eligible provided that they have been treated and CSF is clear for at least 2 weeks prior to enrollment into the study. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Karnofsky/Lansky performance status > 50 %
* Adequate organ function as defined below:

  * Total bilirubin < 2 mg/dL
  * AST(SGOT)/ALT(SGPT) < 3.0 x upper limit of normal (ULN)
  * Creatinine within normal institutional limits OR creatinine clearance > 50 mL/min/1.73 m2 by Schwartz formula or GFR (See Appendix B)
  * Oxygen saturation ≥90% on room air
  * Ejection fraction ≥35%
* Able to be off corticosteroids and any other immune suppressive medications beginning on Day -3 and continuing until 30 days after the infusion of the CIML NK cells. However, use of low-level corticosteroids is permitted if deemed medically necessary. Low-level corticosteroid use is defined as 10mg or less of prednisone (or equivalent for other steroids) per day.
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study and throughout the DLT evaluation period.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Relapsed after allogeneic transplantation.
* Isolated extramedullary relapse
* Circulating blast count >30,000/µL by morphology or flow cytometry (cytoreductive therapies including leukapheresis or hydroxyurea are allowed).
* Patients with any of the following diagnoses:

  * Down's syndrome
  * Acute promyelocytic leukemia (APL)
  * Juvenile myelomonocytic leukemia (JMML)
* Uncontrolled bacterial or viral infections, or known HIV, Hepatitis B or C infection.
* Known hypersensitivity to one or more of the study agents.
* Received any investigational drugs within the 14 days prior to the first dose of fludarabine.
* Pregnant

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (complete remission (CR) plus complete remission with incomplete blood count recovery (CRi)) | Day 28
  * Complete remission (CR) requires all of the following:
    * Bone marrow:
    * Morphologically leukemia free state (≤ 5% myeloblasts) with normal maturation of all cell lines. Persistent dysplasia may be noted
    * Peripheral blood:
    * Platelets ≥ 100,000/uL
    * Neutrophils ≥ 1000/uL
  * Complete remission with incomplete blood count recovery (CRi):
    * All of the above criteria for CR must be met, except that absolute neutrophils <1000/μL or platelets <100,000 /μL in the blood.
Percentage of patients able to proceed to stem cell transplant | Up to 60 days

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 2 years
  -DFS is defined as the time from the day CR or CRi is documented until disease progression or death.
Overall survival (OS) | Up to 2 years
  -OS is defined from the date of first dose of fludarabine on this study until death.
Percentage of patients who achieve minimum residual disease (MRD)-negative status | Day 28
Safety of regimen as measured by number of adverse events | From Day 0 to Day 100
  -Adverse events will be collected from Day 0 to Day 35; however, bone marrow suppression (ANC ≤ 500/mcL) and adverse events of GVHD involving the liver, skin, or gastrointestinal tract will be recorded to Day 100
Duration of remission | Up to 2 years
Time to progression | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bednarski, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu